CLINICAL TRIAL: NCT04494256
Title: A Phase 1/2 Multiple-Ascending-Dose Study With a Long-Term Open-Label Extension to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Effect on Disease Progression of BIIB105 Administered Intrathecally to Adults With Amyotrophic Lateral Sclerosis With or Without Poly-CAG Expansion in the ATXN2 Gene
Brief Title: A Study to Assess the Safety, Tolerability, and Effect on Disease Progression of BIIB105 in Participants With Amyotrophic Lateral Sclerosis (ALS) and Participants With the ALS Ataxin-2 (ATXN2) Genetic Mutation
Acronym: ALSpire
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 275AS101; 2020-000207-36 (EudraCT Number)
Record Dates: First submitted 2020-07-30; First posted 2020-07-31 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1: Cohort A (Experimental): Participants with ALS will receive BIIB105 Dose 1, intrathecally (IT), as 3 loading doses on Day 1 and two later days, followed by two maintenance doses on two later days.
  Interventions: Drug: BIIB105
- Part 1: Cohort B (Experimental): Participants with ALS will receive BIIB105 Dose 2, IT, as 3 loading doses on Day 1 and two later days, followed by two maintenance doses on two later days.
  Interventions: Drug: BIIB105
- Part 1: Cohort C1 (Experimental): Participants with ALS will receive BIIB105 Dose 3, IT, as 3 loading doses on Day 1 and two later days, followed by two maintenance doses on two later days.
  Interventions: Drug: BIIB105
- Part 1: Cohort D1 (Experimental): Participants with ALS will receive BIIB105 Dose 4, IT, as 3 loading doses on Day 1 and two later days, followed by five maintenance doses on five later days.
  Interventions: Drug: BIIB105
- Part 1: Cohort C2 (Experimental): Participants with polyQ-ALS will receive BIIB105 Dose 3, IT, as 3 loading doses on Day 1 and two later days, followed by two maintenance doses on two later days.
  Interventions: Drug: BIIB105
- Part 1: Cohort D2 (Experimental): Participants with polyQ-ALS will receive BIIB105 Dose 4, IT, as 3 loading doses on Day 1 and two later days, followed by five maintenance doses on five later days.
  Interventions: Drug: BIIB105
- Part 1: Cohorts A-D2: Placebo (Placebo Comparator): Participants with ALS and polyQ-ALS for Cohorts A, B, C1 and C2 will receive matching placebo to BIIB105 as 3 loading doses on Day 1 and two later days, followed by two maintenance doses on two later days, and participants with ALS and polyQ-ALS for Cohorts D1 and D2 will receive matching placebo to BIIB105 as 3 loading doses on Day 1 and two later days, followed by five maintenance doses on five later days.
  Interventions: Drug: Placebo
- Part 2: Cohorts A-C2: Open-Label (Experimental): Participants who complete Cohorts A, B, C1, and C2 will receive BIIB105 Dose 3, IT, as 3 loading doses on Day 1 and two later days, followed up to thirty-eight maintenance doses, on up to thirty-eight later days.
  Interventions: Drug: BIIB105
- Part 2: Cohorts D1, D2: Open-Label (Experimental): Participants who complete Cohorts D1 and D2 will have a blinded Loading Dose Period, during which those who received placebo in Part 1 will receive BIIB105 Dose 4, IT, as 3 loading doses on Day 1 and two later days, while those who received BIIB105 in Part 1 will receive 2 loading doses of BIIB105 Dose 4, IT, on Days 1 and one later day, and placebo on Day 15. After the blinded Loading Dose Period, participants will receive BIIB105 Dose 4 up to thirty-eight maintenance doses, on up to thirty-eight later days.
  Interventions: Drug: BIIB105

INTERVENTIONS:
Drug: BIIB105 — Administered as specified in the treatment arm.
  Arms: Part 1: Cohort A; Part 1: Cohort B; Part 1: Cohort C1; Part 1: Cohort C2; Part 1: Cohort D1; Part 1: Cohort D2; Part 2: Cohorts A-C2: Open-Label; Part 2: Cohorts D1, D2: Open-Label
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Part 1: Cohorts A-D2: Placebo

SUMMARY:
The ALSpire Study is a clinical trial evaluating the investigational drug BIIB105 in adults living with amyotrophic lateral sclerosis (ALS).

The ALSpire Study consists of two parts:

* Part 1: 6-month placebo-controlled study. During Part 1, participants are randomly assigned to receive either BIIB105 or placebo in a 3:1 or 2:1 ratio (depending on the participant's assigned Cohort).
* Part 2: up to 3-year long-term open-label extension. During Part 2, all participants receive BIIB105.

The objectives of the study are to evaluate:

* The safety and tolerability of BIIB105 in people with ALS
* What the body does to BIIB105 (also called "pharmacokinetics")
* What BIIB105 does to the body (also called "pharmacodynamics")
* Whether BIIB105 can slow the worsening of clinical function

DETAILED DESCRIPTION:
About BIIB105:

- BIIB105 is an investigational drug designed to reduce the levels of a protein called ATXN2. It is administered intrathecally (via a procedure called lumbar puncture).

ELIGIBILITY:
Key Inclusion Criteria:

Part 1:

* Ability of the participant to understand the purpose and risks of the study and indicate informed consent, and the ability of the participant or the participant's legally authorized representative, to provide signed and dated informed consent and authorization to use protected health information in accordance with national and local privacy regulations.
* No known presence or family history of mutations in the superoxide dismutase 1 (SOD1) or fused in sarcoma (FUS) genes.
* Participants in Cohorts A, B, C1 and D1, must meet the laboratory-supported probable, probable, or definite criteria for diagnosing ALS according to the World Federation of Neurology El Escorial criteria (revised according to the Airlie House Conference 1998 [Brooks 2000]). Participants in Cohort C2 and D2, must meet any of the prior conditions, but may also only meet clinically possible criteria for diagnosing ALS, or exhibit weakness attributable to ALS in the presence of ataxin-2 protein (ATXN2) intermediate repeats.
* In participants in Cohorts C2 and D2, confirmed intermediate cytosine-adenine-guanine/cytosine-adenine-adenine (CAG/CAA) repeat expansion in the ataxin-2 (ATXN2) gene as defined by at least 1 allele carrying 30 to 33 CAG/CAA repeats.
* Slow vital capacity (SVC) criteria:
* In participants in Cohorts A, B, C1, and D1, SVC ≥60% of predicted value as adjusted for sex, age, and height (from the sitting position).
* In participants in Cohort C2 and D2, SVC ≥50% of predicted value as adjusted for sex, age, and height (from the sitting position).
* If taking riluzole, participant must be on a stable dose for ≥30 days prior to Day 1 and expected to remain at that dose until the final study visit, unless the Investigator determines that it should be discontinued for medical reasons, in which case it may not be restarted during the study.
* Participants taking concomitant edaravone at study entry must be on a stable dose for ≥60 days prior to the first dose of study treatment (Day 1). Participants taking concomitant edaravone must be willing to continue with the same dose regimen throughout the study, unless the Investigator determines that edaravone should be discontinued for medical reasons, in which case it may not be restarted during the study. Edaravone may not be administered on dosing days of this study.
* Screening values of coagulation parameters including platelet count, international normalized ratio (INR), prothrombin time (PT), and activated partial thromboplastin time (aPTT) should be within normal ranges.
* Has an informant/caregiver who, in the Investigator's judgment, has frequent and sufficient contact with the participant as to be able to provide accurate information about the participant's cognitive and functional abilities at screening.

Part 2:

* Ability of the participant to understand the purpose and risks of the study and indicate informed consent, and the ability of the participant or the participant's legally authorized representative to provide signed and dated informed consent and authorization to use protected health information in accordance with national and local privacy regulations
* Participants must have completed Study NCT04494256 Part 1 through Week 25 (Day 175 Visit for Cohorts A, B, C1, C2; Day 176 Visit for Cohorts D1, D2). This inclusion criterion does not apply to a participant if Part 1 was terminated by the Sponsor before the participant reached Week 25.
* Participants from Cohorts A, B, C1, and C2 must have a washout of ≥16 weeks between the last dose of study treatment received in Study NCT04494256 Part 1 and the first dose of BIIB105 received in Study NCT04494256 Part 2. Participants from Cohorts D1 and D2 do not require a washout period.
* If taking riluzole, participant must be on a stable dose for ≥30 days prior to Day 1 and expected to remain at that dose until the final study visit, unless the Investigator determines that it should be discontinued for medical reasons, in which case it may not be restarted during the study.
* Participants taking concomitant edaravone at study entry must be on a stable dose for ≥60 days prior to the first dose of study treatment (Day 1). Participants taking concomitant edaravone must be willing to continue with the same dose regimen throughout the study, unless the Investigator determines that edaravone should be discontinued for medical reasons, in which case it may not be restarted during the study. Edaravone may not be administered on dosing days of this study.
* Screening values of coagulation parameters including platelet count, INR, PT, and aPTT should be within normal ranges.

Key Exclusion Criteria

Part 1:

* History or positive test result at Screening for human immunodeficiency virus (HIV).
* Current hepatitis C infection.
* Current hepatitis B infection.
* History of alcohol or substance abuse ≤6 months of Screening that would limit participation in the study, as determined by the Investigator.
* Current or anticipated need, in the opinion of the Investigator, of a diaphragm pacing system during the study period.
* Presence of tracheostomy.
* In participants from Cohorts A, B, C1, and D1, history of myocardial infarction, as determined by the Investigator.
* In participants from Cohorts A, B, C1, and D1, poorly controlled type 1 or 2 diabetes mellitus defined as hemoglobin A1c (HbA1c) ≥8% during Screening.
* In participants in Cohorts A, B, and C1, prescreening ALSFRS-R slope >-0.4 points/month, where prescreening ALSFRS-R slope is defined as: (ALSFRS-R score at Screening - 48) / (months from date of symptom onset to date of Screening). This criterion is not applicable for Cohorts C2, D1, and D2.
* Treatment with another investigational drug (including investigational drugs for ALS through compassionate use programs) or biological agent within 1 month or 5 half-lives of study agent, whichever is longer, before Screening.
* Treatment with an approved disease-modifying therapy for ALS other than riluzole or edaravone within 1 month or 5 half-lives of therapy, whichever is longer, before completion of screening.
* Treatment with an antiplatelet or anticoagulant therapy that cannot safely be interrupted for lumbar puncture (LP) according to local standard of care and/or institutional guidelines, in the opinion of the Investigator or Prescriber.
* Female participants who are pregnant or currently breastfeeding and those intending to become pregnant during the study.

Part 2:

* History or positive test result at Screening for HIV. If participants from Cohorts D1 and D2 who would seamlessly roll from Part 1 into Part 2 test positive for HIV during screening for Part 2 but are clinically asymptomatic, they may enroll in Part 2 at the discretion of the Investigator.
* Current hepatitis C infection. If participants from Cohorts D1 and D2 who would seamlessly roll from Part 1 into Part 2 test positive for hepatitis C during screening for Part 2 but are clinically asymptomatic, they may enroll in Part 2 at the discretion of the Investigator.
* Current hepatitis B infection. If participants from Cohorts D1 and D2 who would seamlessly roll from Part 1 into Part 2 test positive for hepatitis B during screening for Part 2 but are clinically asymptomatic, they may enroll in Part 2 at the discretion of the Investigator.
* History of alcohol or substance abuse ≤ 6 months of Screening that would limit participation in the study, as determined by the Investigator.
* Current or anticipated need, in the opinion of the Investigator, of a diaphragm pacing system during the study period.
* In participants from Cohorts A, B, C1, and D1, history of myocardial infarction, as determined by the Investigator.
* In participants from Cohorts A, B, C1, and D1, poorly controlled type 1 or 2 diabetes mellitus defined as HbA1c ≥8% during Screening.
* Treatment with another investigational drug (including investigational drugs for ALS through compassionate use programs; excluding BIIB105) or biological agent within 1 month or 5 half-lives of study agent, whichever is longer, before Screening.
* Treatment with an antiplatelet or anticoagulant therapy that cannot safely be interrupted for LP according to local standard of care and/or institutional guidelines, in the opinion of the Investigator or Prescriber.
* Female participants who are pregnant or currently breastfeeding and those intending to become pregnant during the study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (17):
- United States (14):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California San Diego Medical Center, La Jolla, California
  - Stanford Neuromuscular Research Center, Palo Alto, California
  - University of Colorado Hospital - Neuroscience Center -Anschutz Medical Campus, Aurora, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Mayo Clinic Florida, Jacksonville, Florida
  - Orlando Health, Orlando, Florida
  - The Emory Clinic, Atlanta, Georgia
  - ALS Clinic - Department of Neurology, Neuromuscular Division, Johns Hopkins University, School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, School of Medicine, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Houston Methodist Neurological Institute, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Montreal Neurological Institute-Hospital, Montreal, Quebec, Canada
- A.O.U. Città della salute e della scienza di Torino, Torino, Italy
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Kim G, Nakayama L, Blum JA, Akiyama T, Boeynaems S, Chakraborty M, Couthouis J, Tassoni-Tsuchida E, Rodriguez CM, Bassik MC, Gitler AD. Genome-wide CRISPR screen reveals v-ATPase as a drug target to lower levels of ALS protein ataxin-2. Cell Rep. 2022 Oct 25;41(4):111508. doi: 10.1016/j.celrep.2022.111508. PMID 36288714
- See also: Biogen Trial Link — https://www.biogentriallink.com/en-us/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with amyotrophic lateral sclerosis (ALS) and ALS associated with ataxin-2 (ATXN2) polyCAG expansion (polyQALS) took part in the study at investigational sites in the United States, Netherlands, Canada and Italy from 28 September 2020 to 13 August 2024.
Pre-assignment Details: A total of 99 participants were randomized in Part 1 (placebo-controlled) of study to receive BIIB105 or placebo, of which 80 participants completed Part 1. A total of 70 eligible participants who completed Part 1 were enrolled into Part 2 (open-label) of study to receive BIIB105. Part 2 of study was terminated early based on Sponsor's decision.
Groups:
- Part 1: Pooled Placebo 1+2: Participants with ALS and polyQ-ALS from Cohorts A, B, C1 and C2 received 3 loading doses of BIIB105-matched placebo, administered every 2 weeks (on Days 1, 15 and 29), followed by 2 maintenance doses administered once every 4 weeks (on Days 57 and 85), for a total of 5 doses over approximately 13 weeks. Participants with ALS and polyQ-ALS from Cohorts D1 and D2 received 3 loading doses of BIIB105- matched placebo administered every 2 weeks (on Days 1, 15, and 29), followed by 5 maintenance doses administered once every 4 weeks (on Days 57, 85, 113, 141, and 169), for a total of 8 doses over approximately 25 weeks.
- Part 1: Cohort A: BIIB105 5 Milligrams (mg): Participants with ALS received 3 loading doses of BIIB105 5mg, intrathecally (IT), administered every 2 weeks (on Days 1, 15, and 29), followed by 2 maintenance doses administered once every 4 weeks (on Days 57 and 85), for a total of 5 doses over approximately 13 weeks.
- Part 1: Cohort B: BIIB105 20 mg: Participants with ALS received 3 loading doses of BIIB105 20mg, IT, administered every 2 weeks (on Days 1, 15, and 29), followed by 2 maintenance doses administered once every 4 weeks (on Days 57 and 85), for a total of 5 doses over approximately 13 weeks.
- Part 1: Cohorts C1+C2: BIIB105 60 mg: Participants with ALS (Cohort C1) and polyQ-ALS (Cohort C2) received 3 loading doses of BIIB105 60 mg, IT, administered every 2 weeks (on Days 1, 15, and 29), followed by 2 maintenance doses administered once every 4 weeks (on Days 57 and 85), for a total of 5 doses over approximately 13 weeks.
- Part 1: Cohorts D1 + D2: BIIB105 120 mg: Participants with ALS (Cohort D1) and polyQ-ALS (Cohort D2) received 3 loading doses of BIIB105 120 mg, IT, administered every 2 weeks (on Days 1, 15, and 29), followed by 5 maintenance doses administered once every 4 weeks (on Days 57, 85, 113, 141, and 169), for a total of 8 doses over approximately 25 weeks.
- Part 2: BIIB105 60 mg: Participants from cohorts A-C2, who received 5, 20 and 60 mg doses of BIIB105 and placebo in Part 1 and completed Week 25 (Day 175) visit in Part 1 received BIIB105 60 mg in Part 2.
- Part 2: BIIB105 120 mg: Participants from Cohorts D1 and D2 who received 120 mg dose of BIIB105 and placebo in Part 1 and completed Week 25 (Day 176) visit in Part 1 received BIIB105 120 mg in Part 2.
Period: Part 1: Double Blinded Period
Arm/Group | Part 1: Pooled Placebo 1+2 | Part 1: Cohort A: BIIB105 5 Milligrams (mg) | Part 1: Cohort B: BIIB105 20 mg | Part 1: Cohorts C1+C2: BIIB105 60 mg | Part 1: Cohorts D1 + D2: BIIB105 120 mg | Part 2: BIIB105 60 mg | Part 2: BIIB105 120 mg
Started | 28 | 6 | 6 | 11 | 48 | 0 | 0
Completed | 26 | 6 | 5 | 9 | 34 | 0 | 0
Not Completed | 2 | 0 | 1 | 2 | 14 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Disease Progression - As Defined by the Protocol | 0 | 0 | 0 | 0 | 5 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — SubjectWithdrawal-VisitBurden/SchedulingConflict | 0 | 0 | 0 | 1 | 3 | 0 | 0
Not completed — Withdrawal by Subject - Other | 1 | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Part 2: Open Label Period
Arm/Group | Part 1: Pooled Placebo 1+2 | Part 1: Cohort A: BIIB105 5 Milligrams (mg) | Part 1: Cohort B: BIIB105 20 mg | Part 1: Cohorts C1+C2: BIIB105 60 mg | Part 1: Cohorts D1 + D2: BIIB105 120 mg | Part 2: BIIB105 60 mg | Part 2: BIIB105 120 mg
Started (Not all participants that completed Part 1 started Part 2.) | 0 | 0 | 0 | 0 | 0 | 19 | 51
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 19 | 51
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 4 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Disease Progression - As Defined by the Protocol | 0 | 0 | 0 | 0 | 0 | 5 | 6
Not completed — Lack of Efficacy - Based on Subject Perception | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 4 | 35
Not completed — SubjectWithdrawal-VisitBurden/SchedulingConflict | 0 | 0 | 0 | 0 | 0 | 5 | 4
Not completed — Withdrawal by Subject - Other | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The part 1 full analysis set (FAS) population included all randomized participants who received at least 1 dose of study treatment in Part 1.
Groups:
- Part 1: Cohort A: BIIB105 5 mg: Participants with ALS received 3 loading doses of BIIB105 5 mg, IT, administered every 2 weeks (on Days 1, 15, and 29), followed by 2 maintenance doses administered once every 4 weeks (on Days 57 and 85), for a total of 5 doses over approximately 13 weeks.
- Part 1: Cohort B: BIIB105 20 mg: Participants with ALS received 3 loading doses of BIIB105 20 mg, IT, administered every 2 weeks (on Days 1, 15, and 29), followed by 2 maintenance doses administered once every 4 weeks (on Days 57 and 85), for a total of 5 doses over approximately 13 weeks.
- Total: Total of all reporting groups
Arm/Group | Part 1: Pooled Placebo 1+2 | Part 1: Cohort A: BIIB105 5 mg | Part 1: Cohort B: BIIB105 20 mg | Part 1: Cohorts C1+C2: BIIB105 60 mg | Part 1: Cohorts D1 + D2: BIIB105 120 mg | Total
Number analyzed (Participants) | 28 | 6 | 6 | 11 | 48 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (11.15) | 60.5 (5.72) | 49.3 (17.84) | 53.3 (12.77) | 57.7 (11.45) | 57.5 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 3 | 3 | 14 | 31
  Male | 19 | 4 | 3 | 8 | 34 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 2 | 1 | 3 | 10
  Not Hispanic or Latino | 23 | 6 | 4 | 10 | 45 | 88
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 3 | 0 | 0 | 0 | 1 | 4
  Black or African American | 0 | 00 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  White | 22 | 6 | 5 | 10 | 40 | 83
  Multiple | 0 | 0 | 0 | 0 | 1 | 1
  Not reported due to confidentiality regulations | 1 | 0 | 0 | 0 | 0 | 1
  Other | 2 | 0 | 1 | 1 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An SAE was any untoward medical occurrence that at any dose results in death, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, or is a medically important event. A TEAE/TESAE was defined as any AE/SAE with an onset date that is on or after the first dose of study drug or any pre-existing condition that has worsened in severity after the first dose of study drug.
Time Frame: From first dose of the study drug in Part 1 up to end of follow up period in Part 1 (up to Day 260)
Population: Part 1 safety analysis population included all randomized participants who received at least 1 dose of study treatment in Part 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Pooled Placebo 1+2 | Part 1: Cohort A: BIIB105 5 mg | Part 1: Cohort B: BIIB105 20 mg | Part 1: Cohorts C1+C2: BIIB105 60 mg | Part 1: Cohorts D1 + D2: BIIB105 120 mg
Number analyzed (Participants) | 28 | 6 | 6 | 11 | 48
Participants
  TEAEs | 28 | 6 | 6 | 11 | 48
  TESAEs | 5 | 0 | 0 | 1 | 7

2. Primary Outcome: Part 2: Number of Participants With TEAEs and TESAEs
Description: as for outcome 1
Time Frame: From first dose of the study in Part 2 up to end of follow up period in Part 2 (up to Day 1184)
Population: Part 2 safety analysis population included all randomized participants who received at least 1 dose of study treatment in Part 2.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: BIIB105 60 mg: Participants from cohorts A-C2, who received 5, 20 and 60 mg BIIB105 and placebo in Part 1 and completed Week 25 (Day 175) Visit in Part 1 received BIIB105 60 mg in Part 2.
- Part 2: BIIB105 120 mg: Participants from Cohorts D1 and D2 randomised to BIIB105 120 mg and placebo in Part 1 and completed Week 25 (Day 176) Visit in Part 1 received BIIB105 at 120 mg in Part 2.
Arm/Group | Part 2: BIIB105 60 mg | Part 2: BIIB105 120 mg
Number analyzed (Participants) | 19 | 51
Participants
  TEAEs | 19 | 49
  TESAEs | 7 | 14

3. Secondary Outcome: Part 1: Serum Concentrations of BIIB105
Time Frame: Pre-dose and 1, 2, 4, 6 hours post-dose on days 1, 15, 29, 57, 85,113, 141, 169 and on days 2, 8, 92, and 176
Population: The Part 1 pharmacokinetic (PK) analysis population included all randomized participants who received at least 1 dose of study treatment and had at least 1 postdose serum and/or cerebrospinal fluid (CSF) BIIB105 measurement in Part 1. 'Number analyzed (n)' signifies number of participants evaluable for this outcome measure (OM) at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part 1: Cohort A: BIIB105 5 mg | Part 1: Cohort B: BIIB105 20 mg | Part 1: Cohorts C1+C2: BIIB105 60 mg | Part 1: Cohorts D1 + D2: BIIB105 120 mg
Number analyzed (Participants) | 6 | 6 | 11 | 48
nanograms per milliliter (ng/mL)
  Day 1: Pre-dose: number analyzed (Participants) | 6 | 6 | 11 | 47
  Day 1: Pre-dose | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 1: 1 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 47
  Day 1: 1 HR post-dose | 7.21 (500.18) | 57.70 (285.30) | 34.98 (465.78) | 187.14 (351.05)
  Day 1: 2 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 47
  Day 1: 2 HR post-dose | 32.20 (177.01) | 135.71 (109.27) | 250.28 (101.57) | 620.38 (132.37)
  Day 1: 4 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 47
  Day 1: 4 HR post-dose | 41.38 (125.95) | 211.34 (68.29) | 488.11 (51.22) | 798.21 (86.03)
  Day 1: 6 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 47
  Day 1: 6 HR post-dose | 39.27 (102.97) | 165.05 (60.63) | 528.45 (61.49) | 774.73 (60.51)
  Day 2 | 6.76 (65.90) | 29.07 (76.82) | 118.70 (103.89) | 260.03 (67.59)
  Day 8: number analyzed (Participants) | 6 | 6 | 11 | 44
  Day 8 | 0.46 (18.74) | 0.47 (36.02) | 1.38 (74.15) | 2.97 (43.60)
  Day 15: Pre-dose: number analyzed (Participants) | 6 | 6 | 11 | 44
  Day 15: Pre-dose | 0.00 (0.00) | 0.50 (20.12) | 0.78 (52.94) | 1.90 (43.15)
  Day 15: 1 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 41
  Day 15: 1 HR post-dose | 3.85 (172.70) | 22.24 (226.26) | 56.01 (489.04) | 257.73 (290.21)
  Day 15: 2 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 41
  Day 15: 2 HR post-dose | 16.89 (111.49) | 94.51 (140.45) | 246.73 (142.61) | 972.44 (110.25)
  Day 15: 4 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 41
  Day 15: 4 HR post-dose | 30.07 (74.48) | 139.75 (137.49) | 363.86 (77.37) | 996.20 (83.48)
  Day 15: 6 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 41
  Day 15: 6 HR post-dose | 27.28 (106.96) | 139.00 (98.33) | 411.61 (49.33) | 897.25 (78.56)
  Day 29: Pre-dose: number analyzed (Participants) | 6 | 6 | 11 | 43
  Day 29: Pre-dose | 0.45 (24.48) | 0.48 (28.47) | 1.23 (64.84) | 2.59 (59.99)
  Day 29: 1 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 42
  Day 29: 1 HR post-dose | 5.80 (117.90) | 16.45 (557.48) | 114.69 (226.87) | 248.00 (152.63)
  Day 29: 2 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 42
  Day 29: 2 HR post-dose | 16.53 (121.68) | 51.58 (602.03) | 420.39 (116.92) | 773.11 (95.92)
  Day 29: 4 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 42
  Day 29: 4 HR post-dose | 31.29 (120.91) | 102.80 (200.28) | 566.43 (71.83) | 953.50 (80.75)
  Day 29: 6 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 40
  Day 29: 6 HR post-dose | 33.28 (127.43) | 151.47 (87.99) | 555.65 (52.83) | 942.06 (69.00)
  Day 57: Pre-dose: number analyzed (Participants) | 6 | 6 | 11 | 41
  Day 57: Pre-dose | 0.00 (0.00) | 0.41 (21.53) | 0.79 (80.26) | 1.83 (69.80)
  Day 57: 1 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 41
  Day 57: 1 HR post-dose | 7.45 (275.61) | 7.98 (159.54) | 44.33 (615.14) | 227.06 (214.59)
  Day 57: 2 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 40
  Day 57: 2 HR post-dose | 22.05 (153.51) | 26.59 (107.62) | 274.02 (128.39) | 713.36 (122.48)
  Day 57: 4 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 41
  Day 57: 4 HR post-dose | 27.72 (123.67) | 74.60 (85.53) | 471.12 (95.76) | 887.82 (105.32)
  Day 57: 6 HR post-dose: number analyzed (Participants) | 6 | 6 | 11 | 40
  Day 57: 6 HR post-dose | 27.33 (105.30) | 89.38 (74.82) | 416.91 (94.12) | 889.54 (89.20)
  Day 85: Pre-dose: number analyzed (Participants) | 6 | 5 | 10 | 41
  Day 85: Pre-dose | 0.50 (0.00) | 0.40 (33.26) | 0.74 (64.453) | 1.91 (113.18)
  Day 85: 1 HR post-dose: number analyzed (Participants) | 6 | 5 | 10 | 40
  Day 85: 1 HR post-dose | 7.02 (111.81) | 18.91 (240.40) | 77.63 (142.75) | 231.31 (236.91)
  Day 85: 2 HR post-dose: number analyzed (Participants) | 6 | 5 | 10 | 40
  Day 85: 2 HR post-dose | 20.60 (95.33) | 69.04 (265.82) | 248.33 (84.14) | 651.00 (127.92)
  Day 85: 4 HR post-dose: number analyzed (Participants) | 6 | 5 | 10 | 40
  Day 85: 4 HR post-dose | 27.69 (111.28) | 140.04 (91.00) | 416.74 (80.90) | 799.70 (89.26)
  Day 85: 6 HR post-dose: number analyzed (Participants) | 6 | 5 | 10 | 40
  Day 85: 6 HR post-dose | 29.83 (119.17) | 140.74 (50.95) | 453.58 (74.39) | 837.50 (73.65)
  Day 92: number analyzed (Participants) | 6 | 5 | 10 | 6
  Day 92 | 0.43 (23.54) | 0.56 (47.98) | 2.05 (92.02) | 4.47 (64.10)
  Day 113: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 39
  Day 113: Pre-dose |  |  |  | 1.95 (59.79)
  Day 113: 1 HR post-dose: number analyzed (Participants) | 0 | 0 | 0 | 39
  Day 113: 1 HR post-dose |  |  |  | 193.04 (198.68)
  Day 113: 2 HR post-dose: number analyzed (Participants) | 0 | 0 | 0 | 39
  Day 113: 2 HR post-dose |  |  |  | 632.28 (91.07)
  Day 113: 4 HR post-dose: number analyzed (Participants) | 0 | 0 | 0 | 39
  Day 113: 4 HR post-dose |  |  |  | 802.46 (91.76)
  Day 113: 6 HR post-dose: number analyzed (Participants) | 0 | 0 | 0 | 39
  Day 113: 6 HR post-dose |  |  |  | 858.58 (86.76)
  Day 141: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 38
  Day 141: Pre-dose |  |  |  | 2.07 (80.82)
  Day 141: 1 HR post-dose: number analyzed (Participants) | 0 | 0 | 0 | 37
  Day 141: 1 HR post-dose |  |  |  | 457.25 (162.57)
  Day 141: 2 HR post-dose: number analyzed (Participants) | 0 | 0 | 0 | 37
  Day 141: 2 HR post-dose |  |  |  | 949.31 (120.40)
  Day 141: 4 HR post-dose: number analyzed (Participants) | 0 | 0 | 0 | 37
  Day 141: 4 HR post-dose |  |  |  | 1044.80 (101.09)
  Day 141: 6 HR post-dose: number analyzed (Participants) | 0 | 0 | 0 | 36
  Day 141: 6 HR post-dose |  |  |  | 996.44 (85.54)
  Day 169: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 36
  Day 169: Pre-dose |  |  |  | 2.95 (153.02)
  Day 169: 1 HR post-dose: number analyzed (Participants) | 0 | 0 | 0 | 35
  Day 169: 1 HR post-dose |  |  |  | 288.75 (217.19)
  Day 169: 2 HR post-dose: number analyzed (Participants) | 0 | 0 | 0 | 35
  Day 169: 2 HR post-dose |  |  |  | 702.24 (107.10)
  Day 169: 4 HR post-dose: number analyzed (Participants) | 0 | 0 | 0 | 36
  Day 169: 4 HR post-dose |  |  |  | 816.90 (86.61)
  Day 169: 6 HR post-dose: number analyzed (Participants) | 0 | 0 | 0 | 37
  Day 169: 6 HR post-dose |  |  |  | 683.89 (158.85)
  Day 176: number analyzed (Participants) | 0 | 0 | 0 | 33
  Day 176 |  |  |  | 6.97 (132.41)

4. Secondary Outcome: Part 1: CSF Concentrations of BIIB105
Time Frame: Pre-dose on Days 1, 15, 29, 57, 85, 113, 141, 169, and on days 92, 130, 175, and 176
Population: The Part 1 PK analysis population included all randomized participants who received at least 1 dose of study treatment and had at least 1 postdose serum and/or CSF BIIB105 measurement in Part 1. 'Number analyzed (n)' signifies number of participants evaluable for this OM at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Cohort A: BIIB105 5 mg | Part 1: Cohort B: BIIB105 20 mg | Part 1: Cohorts C1+C2: BIIB105 60 mg | Part 1: Cohorts D1 + D2: BIIB105 120 mg
Number analyzed (Participants) | 6 | 6 | 11 | 48
ng/mL
  Day 1 : Pre-dose: number analyzed (Participants) | 6 | 6 | 11 | 47
  Day 1 : Pre-dose | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 15 : Pre-dose: number analyzed (Participants) | 6 | 6 | 11 | 44
  Day 15 : Pre-dose | 1.93 (41.54) | 2.71 (55.21) | 5.75 (62.33) | 14.54 (82.48)
  Day 29 : Pre-dose: number analyzed (Participants) | 6 | 6 | 11 | 43
  Day 29 : Pre-dose | 3.53 (33.52) | 4.32 (52.42) | 11.53 (49.38) | 17.53 (95.18)
  Day 57 : Pre-dose: number analyzed (Participants) | 6 | 6 | 11 | 42
  Day 57 : Pre-dose | 2.32 (28.96) | 2.65 (46.23) | 4.82 (59.33) | 10.29 (79.90)
  Day 85 : Pre-dose: number analyzed (Participants) | 6 | 5 | 10 | 40
  Day 85 : Pre-dose | 2.37 (30.35) | 3.18 (72.73) | 6.50 (36.23) | 14.06 (77.42)
  Day 92: number analyzed (Participants) | 6 | 5 | 10 | 0
  Day 92 | 5.01 (30.62) | 6.28 (74.45) | 25.51 (66.26) |
  Day 113: number analyzed (Participants) | 0 | 0 | 0 | 40
  Day 113 |  |  |  | 17.08 (86.41)
  Day 130: number analyzed (Participants) | 6 | 5 | 10 | 0
  Day 130 | 2.09 (32.22) | 2.45 (57.06) | 5.42 (40.72) |
  Day 141: number analyzed (Participants) | 0 | 0 | 0 | 38
  Day 141 |  |  |  | 17.91 (84.83)
  Day 169: number analyzed (Participants) | 0 | 0 | 0 | 37
  Day 169 |  |  |  | 18.88 (74.23)
  Day 175: number analyzed (Participants) | 6 | 6 | 11 | 0
  Day 175 | 1.16 (54.77) | 1.16 (36.06) | 2.68 (46.05) |
  Day 176: number analyzed (Participants) | 0 | 0 | 0 | 2
  Day 176 |  |  |  | 17.35 (0.04)

5. Secondary Outcome: Part 1: Area Under the Serum Concentration-Time Curve From Time Zero to Infinity (AUCinf)
Description: AUCinf is the area under the serum concentration-time profile from time 0 extrapolated to infinite time. AUCinf was reported following dose 1 as planned.
Time Frame: Day 1
Population: Part 1 PK analysis population included all randomized participants who received at least 1 dose of study treatment and had at least 1 postdose serum and/or CSF BIIB105 measurement in Part 1. 'Overall number of participants analyzed' signifies number of participants with data available for OM analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1: Cohort A: BIIB105 5 mg | Part 1: Cohort B: BIIB105 20 mg | Part 1: Cohorts C1+C2: BIIB105 60 mg | Part 1: Cohorts D1 + D2: BIIB105 120 mg
Number analyzed (Participants) | 2 | 5 | 10 | 42
Hour*nanogram per milliliter (h*ng/mL) | 934.22 (52.89) | 3546.89 (53.50) | 11258.45 (14.57) | 24466.44 (30.24)

6. Secondary Outcome: Part 1: Area Under the Serum Concentration-Time Curve From Time Zero to Time of the Last Measurable Concentration (AUClast)
Description: AUClast was reported following dose 1 as planned.
Time Frame: Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: Cohort A: BIIB105 5 mg | Part 1: Cohort B: BIIB105 20 mg | Part 1: Cohorts C1+C2: BIIB105 60 mg | Part 1: Cohorts D1 + D2: BIIB105 120 mg
Number analyzed (Participants) | 6 | 6 | 11 | 44
h*ng/mL | 574.59 (79.16) | 3239.40 (52.73) | 11758.68 (21.12) | 24289.70 (30.50)

7. Secondary Outcome: Part 1: Maximum Observed Serum Concentration (Cmax)
Time Frame: Days 1, 15, 29, 57, 85, 113, 141 and 169
Population: Part 1 PK analysis population included all randomized participants who received at least 1 dose of study treatment and had at least 1 postdose serum and/or CSF BIIB105 measurement in Part 1. 'Number analyzed (n)' signifies number of participants evaluable for this OM at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Cohort A: BIIB105 5 mg | Part 1: Cohort B: BIIB105 20 mg | Part 1: Cohorts C1+C2: BIIB105 60 mg | Part 1: Cohorts D1 + D2: BIIB105 120 mg
Number analyzed (Participants) | 6 | 6 | 11 | 48
ng/mL
  Day 1: number analyzed (Participants) | 6 | 6 | 11 | 47
  Day 1 | 52.18 (123.13) | 227.80 (73.20) | 644.10 (55.31) | 1019.11 (76.61)
  Day 15: number analyzed (Participants) | 6 | 6 | 11 | 41
  Day 15 | 31.03 (78.23) | 165.37 (118.45) | 495.03 (76.73) | 1312.42 (93.96)
  Day 29: number analyzed (Participants) | 6 | 6 | 11 | 40
  Day 29 | 34.11 (119.62) | 164.15 (101.46) | 616.02 (61.54) | 1173.71 (75.74)
  Day 57: number analyzed (Participants) | 6 | 6 | 11 | 40
  Day 57 | 31.92 (136.57) | 94.60 (75.30) | 513.84 (98.01) | 1052.70 (99.57)
  Day 85: number analyzed (Participants) | 6 | 5 | 10 | 40
  Day 85 | 31.43 (117.43) | 168.38 (59.96) | 476.91 (75.87) | 1009.44 (84.68)
  Day 113: number analyzed (Participants) | 0 | 0 | 0 | 39
  Day 113 |  |  |  | 949.58 (83.69)
  Day 141: number analyzed (Participants) | 0 | 0 | 0 | 36
  Day 141 |  |  |  | 1243.75 (91.13)
  Day 169: number analyzed (Participants) | 0 | 0 | 0 | 36
  Day 169 |  |  |  | 957.24 (86.51)

8. Secondary Outcome: Part 1: Time to Reach Maximum Observed Serum Concentration (Tmax)
Time Frame: Days 1, 15, 29, 57, 85, 113, 141 and 169
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: Cohort A: BIIB105 5 mg | Part 1: Cohort B: BIIB105 20 mg | Part 1: Cohorts C1+C2: BIIB105 60 mg | Part 1: Cohorts D1 + D2: BIIB105 120 mg
Number analyzed (Participants) | 6 | 6 | 11 | 48
hour
  Day 1: number analyzed (Participants) | 6 | 6 | 11 | 47
  Day 1 | 4.2 [2 to 6] | 4.2 [2 to 6] | 5.8 [2 to 23] | 4.3 [1 to 24]
  Day 15: number analyzed (Participants) | 6 | 6 | 11 | 41
  Day 15 | 5.0 [4 to 6] | 5.0 [2 to 6] | 5.9 [2 to 6] | 4.1 [1 to 6]
  Day 29: number analyzed (Participants) | 6 | 6 | 11 | 40
  Day 29 | 5.8 [4 to 6] | 5.8 [2 to 6] | 4.2 [2 to 6] | 4.1 [2 to 6]
  Day 57: number analyzed (Participants) | 6 | 6 | 11 | 40
  Day 57 | 5.8 [2 to 6] | 5.0 [4 to 6] | 4.2 [1 to 6] | 4.5 [1 to 6]
  Day 85: number analyzed (Participants) | 6 | 5 | 10 | 40
  Day 85 | 5.1 [4 to 6] | 4.3 [4 to 6] | 5.8 [4 to 6] | 5.8 [2 to 6]
  Day 113: number analyzed (Participants) | 0 | 0 | 0 | 39
  Day 113 |  |  |  | 5.3 [1 to 6]
  Day 141: number analyzed (Participants) | 0 | 0 | 0 | 36
  Day 141 |  |  |  | 4.0 [1 to 6]
  Day 169: number analyzed (Participants) | 0 | 0 | 0 | 36
  Day 169 |  |  |  | 4.1 [1 to 6]

9. Secondary Outcome: Part 1: Elimination Half-Life (t1/2) in Serum
Description: Elimination half-life (t1/2) was reported following dose 1 as planned.
Time Frame: Day 1
Population: Part 1 PK analysis population included all randomized participants who received at least 1 dose of study treatment and had at least 1 postdose serum and/or CSF BIIB105 measurement in Part 1. ''Overall number of participants (n)' signifies number of participants evaluable for this OM.
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: Cohort A: BIIB105 5 mg | Part 1: Cohort B: BIIB105 20 mg | Part 1: Cohorts C1+C2: BIIB105 60 mg | Part 1: Cohorts D1 + D2: BIIB105 120 mg
Number analyzed (Participants) | 2 | 5 | 10 | 42
hour | 14.0 [5 to 23] | 26.6 [17 to 62] | 41.7 [33 to 62] | 39.8 [22 to 82]

10. Secondary Outcome: Part 1: Neurofilament Light Chain (NfL) Plasma Concentration Ratio to Baseline
Description: Plasma NfL ratio to baseline was reported in terms of geometric mean ratio.
Time Frame: Days 29, 57, 85, 113, 130 (For cohorts A, B, C1 and C2)/141 (For cohorts D1 and D2), 169 (For cohorts A, B, C1 and C2)/175 (For cohorts D1 and D2) and 241
Population: The Part 1 pharmacodynamic (PD) population included participants who received at least 1 dose of study treatment and have at least 1 available postdose evaluation of the respective PD endpoint in the study in Part 1. 'Number analyzed (n)' indicates the number of participants evaluable for the OM at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part 1: Pooled Placebo 1+2 | Part 1: Cohort A: BIIB105 5 mg | Part 1: Cohort B: BIIB105 20 mg | Part 1: Cohorts C1+C2: BIIB105 60 mg | Part 1: Cohorts D1 + D2: BIIB105 120 mg
Number analyzed (Participants) | 28 | 6 | 6 | 11 | 47
ratio
  Day 29: number analyzed (Participants) | 28 | 6 | 6 | 11 | 45
  Day 29 | 1.04 (20.32) | 1.05 (8.47) | 0.83 (47.1) | 1.06 (11.23) | 1.15 (72.72)
  Day 57: number analyzed (Participants) | 28 | 6 | 6 | 11 | 44
  Day 57 | 1.08 (19.91) | 0.95 (14.63) | 0.97 (15.95) | 1.08 (20.43) | 1.03 (21.7)
  Day 85: number analyzed (Participants) | 27 | 6 | 5 | 10 | 41
  Day 85 | 0.99 (17.27) | 0.99 (15.7) | 0.98 (26.4) | 1.11 (19.85) | 0.99 (19.62)
  Day 113: number analyzed (Participants) | 17 | 0 | 0 | 0 | 40
  Day 113 | 1.06 (19.95) |  |  |  | 1.01 (21.77)
  Day 130 (A,B,C1,C2)/Day 141 (D1,D2): number analyzed (Participants) | 25 | 6 | 5 | 10 | 39
  Day 130 (A,B,C1,C2)/Day 141 (D1,D2) | 1.09 (20.46) | 1.10 (8.58) | 0.92 (40.79) | 0.99 (30.8) | 1.03 (41.35)
  Day 169 (A,B,C1,C2)/Day 175 (D1,D2): number analyzed (Participants) | 24 | 6 | 5 | 9 | 39
  Day 169 (A,B,C1,C2)/Day 175 (D1,D2) | 1.10 (23.67) | 1.02 (22.58) | 1.10 (24.55) | 1.08 (29.73) | 1.06 (24.92)
  Day 214: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Day 214 |  |  |  |  | 1.07

11. Secondary Outcome: Integrated Part 1 and Part 2: CSF PK Concentration of BIIB105
Time Frame: Predose on Days 1,15,29,57,85 and on Days 1,15,29,57,85,113,141,169.176,197,210,225,253,281,309,337,365,393,420,448,476,504,532,560,588,616,644,672,700,726,728
Population: Integrated Part 1 & 2=Part 1 PK population.Overall number of participants analyzed=number of participants evaluable for OM analysis.Number analyzed=number of participants evaluable at specified timepoint.Assessment was planned upto Day 1093 however,no assessments were conducted after Day 729 due to early termination.Treatment groups for integrated analysis of Parts 1 & 2 were planned for Early-start BIIB105 120 mg & Placebo/Delayed-start BIIB105,& results are reported for these treatment groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Early-start BIIB105 120 mg: Participants from Cohorts D1 and D2 from the Part 1 FAS population who received BIIB105 120 mg in Part 1, who may or may not have continued their study treatment in Part 2 were included in this group.
- Placebo/Delayed-start BIIB105 120 mg: Participants from Cohorts D1 and D2 from the Part 1 FAS population who received placebo in Part 1, who may or may not have rolled over to Part 2 and started active treatment with BIIB105 were included in this group.
Arm/Group | Early-start BIIB105 120 mg | Placebo/Delayed-start BIIB105 120 mg
Number analyzed (Participants) | 48 | 17
ng/mL
  Day 1 : Pre-dose: number analyzed (Participants) | 48 | 0
  Day 1 : Pre-dose | 0.13 (0.00) |
  Day 1: number analyzed (Participants) | 0 | 17
  Day 1 |  | 0.15 (37.88)
  Day 15 : Pre-dose: number analyzed (Participants) | 44 | 0
  Day 15 : Pre-dose | 14.54 (82.48) |
  Day 15: number analyzed (Participants) | 1 | 17
  Day 15 | 31.04 | 12.93 (70.31)
  Day 29: Pre-dose: number analyzed (Participants) | 43 | 0
  Day 29: Pre-dose | 17.53 (95.18) |
  Day 29: number analyzed (Participants) | 0 | 17
  Day 29 |  | 18.62 (93.41)
  Day 57 : Pre-dose: number analyzed (Participants) | 42 | 0
  Day 57 : Pre-dose | 10.29 (79.90) |
  Day 57: number analyzed (Participants) | 0 | 14
  Day 57 |  | 9.72 (49.08)
  Day 85 : Pre-dose: number analyzed (Participants) | 40 | 0
  Day 85 : Pre-dose | 14.06 (77.42) |
  Day 85: number analyzed (Participants) | 0 | 13
  Day 85 |  | 14.54 (63.76)
  Day 113: number analyzed (Participants) | 40 | 11
  Day 113 | 17.08 (86.41) | 20.70 (56.82)
  Day 141: number analyzed (Participants) | 38 | 8
  Day 141 | 17.91 (84.83) | 24.50 (30.13)
  Day 169: number analyzed (Participants) | 37 | 7
  Day 169 | 18.88 (74.23) | 19.32 (36.08)
  Day 176: number analyzed (Participants) | 2 | 0
  Day 176 | 17.35 (0.04) |
  Day 197: number analyzed (Participants) | 32 | 5
  Day 197 | 24.88 (57.69) | 24.99 (71.18)
  Day 210: number analyzed (Participants) | 31 | 0
  Day 210 | 49.04 (67.88) |
  Day 225: number analyzed (Participants) | 33 | 5
  Day 225 | 24.14 (63.21) | 30.52 (13.97)
  Day 253: number analyzed (Participants) | 33 | 5
  Day 253 | 23.54 (62.86) | 21.68 (70.34)
  Day 281: number analyzed (Participants) | 27 | 2
  Day 281 | 26.51 (73.96) | 23.79 (8.69)
  Day 309: number analyzed (Participants) | 25 | 2
  Day 309 | 27.14 (63.54) | 30.47 (13.01)
  Day 337: number analyzed (Participants) | 20 | 2
  Day 337 | 31.34 (71.84) | 22.11 (16.80)
  Day 365: number analyzed (Participants) | 16 | 0
  Day 365 | 30.16 (62.35) |
  Day 393: number analyzed (Participants) | 11 | 2
  Day 393 | 23.56 (31.29) | 15.36 (13.95)
  Day 420: number analyzed (Participants) | 11 | 1
  Day 420 | 25.84 (42.82) | 21.91
  Day 448: number analyzed (Participants) | 9 | 1
  Day 448 | 23.53 (40.75) | 28.43 (NA) — Geometric coefficient of variation is not estimable due to less number of participants.
  Day 476: number analyzed (Participants) | 7 | 1
  Day 476 | 30.87 (28.29) | 25.95 (NA) — Geometric coefficient of variation is not estimable due to less number of participants.
  Day 504: number analyzed (Participants) | 6 | 0
  Day 504 | 28.24 (38.06) |
  Day 532: number analyzed (Participants) | 5 | 0
  Day 532 | 26.73 (44.19) |
  Day 560: number analyzed (Participants) | 4 | 0
  Day 560 | 26.42 (36.82) |
  Day 588: number analyzed (Participants) | 3 | 0
  Day 588 | 40.26 (68.00) |
  Day 616: number analyzed (Participants) | 3 | 0
  Day 616 | 24.69 (109.22) |
  Day 644: number analyzed (Participants) | 4 | 0
  Day 644 | 21.15 (39.95) |
  Day 672: number analyzed (Participants) | 3 | 0
  Day 672 | 30.75 (48.18) |
  Day 700: number analyzed (Participants) | 2 | 0
  Day 700 | 23.85 (1.63) |
  Day 726: number analyzed (Participants) | 1 | 0
  Day 726 | 28.22 |
  Day 728: number analyzed (Participants) | 1 | 0
  Day 728 | 26.28 |

12. Secondary Outcome: Integrated Part 1 and Part 2: Serum Concentration of BIIB105
Time Frame: Up to Day 176
Population: Assessments were planned upto Day 1009 for this OM;however no assessments were conducted after Day 176 due to early termination.Serum concentrations of BIIB105 were not estimable for Integrated Parts 1 & 2.Data collected for serum PK concentrations for Parts 1 & 2 are reported in OM #3 and #20(post-hoc)respectively.Treatment groups for integrated analysis of Parts 1 & 2 were planned for Early-start BIIB105 120 mg & Placebo/Delayed-start BIIB105,& results are reported for these treatment groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Early-start BIIB105 120 mg | Placebo/Delayed-start BIIB105 120 mg
Number analyzed (Participants) | 48 | 17
ng/mL | NA (NA) — Data were not estimable due to values being below the lower limit of quantification | NA (NA) — Data were not estimable due to values being below the lower limit of quantification

13. Secondary Outcome: Integrated Part 1 and Part 2: Neurofilament Light Chain (NfL) Plasma Concentration Ratio to Baseline
Description: Plasma NfL ratio to baseline was reported in terms of geometric mean ratio.
Time Frame: Days 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, 337, 365, 393, 421, 449, 477, 505, 533, 561, 589, 617, 645, 673, 701
Population: Integrated Parts 1 and 2=Part 1 PD population. Number analyzed indicates the number of participants evaluable for the OM at the specified timepoint. The treatment groups for the integrated analysis of Part 1 and Part 2 were planned for Early-start BIIB105 120 mg and Placebo/Delayed-start BIIB105, and results are reported for these treatment groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Early-start BIIB105 120 mg | Placebo/Delayed-start BIIB105 120 mg
Number analyzed (Participants) | 47 | 19
ratio
  Day 29: number analyzed (Participants) | 45 | 19
  Day 29 | 1.15 (72.72) | 1.03 (22.35)
  Day 57: number analyzed (Participants) | 44 | 19
  Day 57 | 1.03 (21.7) | 1.11 (18.9)
  Day 85: number analyzed (Participants) | 41 | 18
  Day 85 | 0.99 (19.62) | 1.00 (18.00)
  Day 113: number analyzed (Participants) | 40 | 17
  Day 113 | 1.01 (21.77) | 1.06 (19.95)
  Day 141: number analyzed (Participants) | 39 | 16
  Day 141 | 1.03 (41.35) | 1.10 (20.84)
  Day 169: number analyzed (Participants) | 39 | 16
  Day 169 | 1.06 (24.92) | 1.06 (20.33)
  Day 197: number analyzed (Participants) | 31 | 13
  Day 197 | 1.08 (28.28) | 1.08 (23.6)
  Day 225: number analyzed (Participants) | 31 | 13
  Day 225 | 1.12 (38.42) | 1.12 (31.12)
  Day 253: number analyzed (Participants) | 26 | 12
  Day 253 | 1.15 (28.4) | 1.06 (27.71)
  Day 281: number analyzed (Participants) | 22 | 10
  Day 281 | 1.14 (26.57) | 1.18 (21.26)
  Day 309: number analyzed (Participants) | 17 | 9
  Day 309 | 1.07 (31.81) | 1.09 (24.46)
  Day 337: number analyzed (Participants) | 12 | 6
  Day 337 | 1.05 (38.67) | 1.18 (23.3)
  Day 365: number analyzed (Participants) | 11 | 4
  Day 365 | 0.99 (32.42) | 1.20 (29.59)
  Day 393: number analyzed (Participants) | 9 | 4
  Day 393 | 0.95 (48.05) | 1.26 (24.88)
  Day 421: number analyzed (Participants) | 9 | 3
  Day 421 | 0.92 (36.61) | 1.21 (58.82)
  Day 449: number analyzed (Participants) | 7 | 3
  Day 449 | 0.82 (28.9) | 1.06 (32.94)
  Day 477: number analyzed (Participants) | 5 | 2
  Day 477 | 0.85 (23.15) | 0.92 (32.52)
  Day 505: number analyzed (Participants) | 3 | 2
  Day 505 | 0.77 (25.18) | 0.88 (46.94)
  Day 533: number analyzed (Participants) | 4 | 2
  Day 533 | 0.78 (14.58) | 1.15 (32.24)
  Day 561: number analyzed (Participants) | 3 | 0
  Day 561 | 0.65 (14.63) |
  Day 589: number analyzed (Participants) | 3 | 2
  Day 589 | 0.77 (39.28) | 0.90 (23.38)
  Day 617: number analyzed (Participants) | 3 | 1
  Day 617 | 0.80 (38.48) | 0.70
  Day 645: number analyzed (Participants) | 2 | 0
  Day 645 | 0.76 (52.68) |
  Day 673: number analyzed (Participants) | 2 | 0
  Day 673 | 0.66 (30.22) |
  Day 701: number analyzed (Participants) | 1 | 0
  Day 701 | 0.54 |

14. Secondary Outcome: Integrated Part 1 and Part 2: Change From Baseline in Percent Predicted Slow Vital Capacity (SVC)
Description: Vital capacity was measured by means of the slow vital capacity (SVC) test using a facemask with the participant sitting upright. SVC was determined by performing at least 3 trials. If the difference between the two highest values of the three trials was ≥10%, then up to 5 trials were performed. The highest percent predicted SVC value at each visit was used for the analysis. Here, baseline is defined as Part 1 day 1 value prior to the study drug. As specified in SAP, change from baseline at Week 40 (Day 281) in least square means and corresponding standard errors was summarized using the analysis of covariance (ANCOVA) model. Negative change from baseline indicates decrease in lung function.
Time Frame: Baseline, Day 281
Population: Integrated data for Part 1 and Part 2 was analyzed based on the clinical function population defined for Part 1. The Part 1 clinical function population included participants from the FAS population who have at least 1 postdose measurement in Part 1. The treatment groups for the integrated analysis of Part 1 and Part 2 were planned for Early-start BIIB105 120 mg and Placebo/Delayed-start BIIB105, and results are reported for these treatment groups.
Measure: Least Squares Mean (Standard Error); unit: percent predicted
Arm/Group | Early-start BIIB105 120 mg | Placebo/Delayed-start BIIB105 120 mg
Number analyzed (Participants) | 48 | 19
percent predicted | -14.49 (4.093) | -14.41 (7.133)
Statistical Analysis 1: Comparison: Early-start BIIB105 120 mg vs Placebo/Delayed-start BIIB105 120 mg; Test type: Superiority; p = 0.9924, ANCOVA — ANCOVA model included: treatment as a fixed effect and adjusted for the following covariates: baseline disease duration since symptom onset, baseline percent predicted SVC, baseline plasma NfL, and use of riluzole or edaravone; Least square (LS) mean difference = -0.1, 95% CI 2-sided [-15.47 to 15.32], Standard Error of Mean 7.84

15. Secondary Outcome: Integrated Part 1 and Part 2: Change From Baseline in Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) Score
Description: The ALSFRS-R is a questionnaire that measured degree of impairment in 4 functional domains: respiratory function, bulbar function, gross motor skills, and fine motor skills. Each domain consists of 3 items, each scored from 0 to 4, with higher scores representing better function. Each domain score can have maximum score of 12 calculated as the sum of scores of 3 items for that domain and the total possible score for ALSFRS-R is 48. The total score is the sum of the 4 functional domain scores or all individual item scores if no missing item scores are present. Here, baseline is defined as Part 1 day 1 value prior to the study drug Negative change from baseline indicates disease progression. As specified in SAP change from baseline at Week 40 (Day 281) in least square means and corresponding standard errors was summarized using the ANCOVA model.
Time Frame: Baseline, Day 281
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Early-start BIIB105 120 mg | Placebo/Delayed-start BIIB105 120 mg
Number analyzed (Participants) | 48 | 19
score on a scale | -8.46 (1.105) | -8.26 (1.819)
Statistical Analysis 1: Comparison: Early-start BIIB105 120 mg vs Placebo/Delayed-start BIIB105 120 mg; Test type: Superiority; p = 0.9203, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LS mean difference = -0.2, 95% CI 2-sided [-4.14 to 3.74], Standard Error of Mean 2.01

16. Secondary Outcome: Integrated Part 1 and Part 2: Change From Baseline in Muscle Strength as Measured by Handheld Dynamometry (HHD) Megascore
Description: Quantitative muscle strength was evaluated using HHD, which tested the isometric strength of multiple muscles using standard participant positioning. Approximately 8 muscle groups were examined (per each side) in both upper and lower extremities. The muscle strength values were normalized to Z scores as (post-baseline measurements -mean)/SD and averaged to provide HHD overall megascore. The overall megascore was created by averaging Z scores, if no more than 14 (≤ 14) measures are missing. A Z-score (also called a standard score) is a way to describe how far and in what direction a data point is from the mean of the dataset (in this case, positive values indicate strength and negative values indicate weakness). A Z-score of 0 indicates the population mean, and a positive score indicates muscle strength. A negative change from baseline indicated decreased muscle strength.
Time Frame: Baseline, Day 281
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Early-start BIIB105 120 mg | Placebo/Delayed-start BIIB105 120 mg
Number analyzed (Participants) | 48 | 19
z-score | -0.407 (0.3918) | -0.439 (0.4406)
Statistical Analysis 1: Comparison: Early-start BIIB105 120 mg vs Placebo/Delayed-start BIIB105 120 mg; Test type: Superiority; p = 0.1069, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LS mean difference = -0.2, 95% CI 2-sided [-0.41 to 0.04], Standard Error of Mean 0.12

17. Secondary Outcome: Integrated Part 1 and Part 2: Time to Death or Permanent Ventilation
Description: Time to death or permanent ventilation is defined as the time from first dose to death or permanent ventilation ( ≥ 22 hours of mechanical ventilation [invasive or noninvasive] per day for ≥ 21 consecutive days), whichever comes first. Participants who did not meet the endpoint definition were censored on the date of participant's last contact in Part 1 or Part 2. Time to death or permanent ventilation data was summarized using Kaplan-Meier curves based on randomization in Part 1.
Time Frame: Baseline up to Day 1184
Population: Integrated data for Part 1 and Part 2 was analyzed based on the FAS population defined for Part 1. Part 1 FAS population included all randomized participants who received at least 1 dose of study treatment in Part 1 and 2. The treatment groups for the integrated analysis of Part 1 and Part 2 were planned for Early-start BIIB105 120 mg and Placebo/Delayed-start BIIB105, and results are reported for these treatment groups.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Early-start BIIB105 120 mg | Placebo/Delayed-start BIIB105 120 mg
Number analyzed (Participants) | 48 | 19
weeks | NA [72.7 to NA] — Median and 95% confidence interval (CI) were not estimable due to low number events of permanent ventilation or death. | NA [NA to NA] — Median and 95% confidence interval (CI) were not estimable due to low number events of permanent ventilation or death.
Statistical Analysis 1: Comparison: Early-start BIIB105 120 mg vs Placebo/Delayed-start BIIB105 120 mg; Test type: Superiority; p = 0.1003, Log Rank; Log rank test stratified by median baseline plasma NfL; Hazard Ratio (HR) = 4.29, 95% CI 2-sided [0.433 to 42.587]

18. Secondary Outcome: Integrated Parts 1 and 2: Time to Death
Description: Time to death was defined as the time from first dose to death.
Time Frame: Baseline up to Day 1184
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Early-start BIIB105 120 mg | Placebo/Delayed-start BIIB105 120 mg
Number analyzed (Participants) | 48 | 19
weeks | NA [NA to NA] — Median and 95% CI were not estimable due to low number of events of death. | NA [NA to NA] — Median and 95% CI were not estimable due to low number of events of death.
Statistical Analysis 1: Comparison: Early-start BIIB105 120 mg vs Placebo/Delayed-start BIIB105 120 mg; Test type: Superiority; p = 0.1143, Kaplan-Meier product limit method

19. Secondary Outcome: Integrated Part 1 and Part 2: Time to Death, Incorporating Post-Study Withdrawal or Study Completion Vital Status Data
Time Frame: Up to Day 1184
Population: As per the changes to the protocol-specified analyses mentioned in the SAP, time to death, incorporating post-study withdrawal or study completion vital status data was not performed as post-study withdrawal vital status data was not collected at the time of this analysis. The treatment groups for the integrated analysis of Part 1 and Part 2 were planned for Early-start BIIB105 120 mg and Placebo/Delayed-start BIIB105, and results are reported for these treatment groups.
Arm/Group | Early-start BIIB105 120 mg | Placebo/Delayed-start BIIB105 120 mg
Number analyzed (Participants) | 0 | 0

20. Post Hoc Outcome: Part 2: Serum Concentration of BIIB105
Time Frame: Days 1, 169, 337, 505 and 673
Population: The PK analysis population is defined as all randomized participants who received at least 1 dose of study treatment and have at least 1 postdose serum and/or CSF BIIB105 measurement. 'Number analyzed' indicates the number of participants evaluable at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: BIIB105 60 mg | Part 2: BIIB105 120 mg
Number analyzed (Participants) | 19 | 51
ng/mL
  Day 1: number analyzed (Participants) | 19 | 50
  Day 1 | 0.50 (0.00) | 1.47 (139.00)
  Day 169: number analyzed (Participants) | 11 | 18
  Day 169 | 1.25 (186.75) | 3.50 (151.48)
  Day 337: number analyzed (Participants) | 9 | 7
  Day 337 | 2.46 (333.20) | 2.50 (95.95)
  Day 505: number analyzed (Participants) | 7 | 1
  Day 505 | 3.53 (340.11) | 8.54 (0.00)
  Day 673: number analyzed (Participants) | 3 | 0
  Day 673 | 18.89 (164.41) |

ADVERSE EVENTS:
Time Frame: From first dose of the study drug up to end of follow up period in Part 1 (up to Day 260) and Part 2 (up to Day 1184)
Description: The Part 1 safety analysis population included all randomized participants who received at least 1 dose of study treatment in Part 1. The Part 2 safety analysis population included all participants who received at least 1 dose of study treatment in Part 2.
Groups:
- Part 1: Cohort A: BIIB105 5 mg: Participants with ALS received 3 loading doses of BIIB105 5mg, IT, administered every 2 weeks (on Days 1, 15, and 29), followed by 2 maintenance doses administered once every 4 weeks (on Days 57 and 85), for a total of 5 doses over approximately 13 weeks.
- Part 1: Cohorts D1 + D2: BIIB105 120 mg: Participants with ALS (Cohort D1) and polyQ-ALS (Cohort D2) received BIIB105 120 mg, IT, as 3 loading doses administered every 2 weeks (on Days 1, 15, and 29), followed by 5 maintenance doses administered once every 4 weeks (on Days 57, 85, 113, 141, and 169), for a total of 8 doses over approximately 25 weeks.
Arm/Group | Part 1: Pooled Placebo 1+2 | Part 1: Cohort A: BIIB105 5 mg | Part 1: Cohort B: BIIB105 20 mg | Part 1: Cohorts C1+C2: BIIB105 60 mg | Part 1: Cohorts D1 + D2: BIIB105 120 mg | Part 2: BIIB105 60 mg | Part 2: BIIB105 120 mg
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/6 | 0/6 | 0/11 | 0/48 | 4/19 | 2/51
Serious Adverse Events (participants affected / at risk) | 5/28 | 0/6 | 0/6 | 1/11 | 7/48 | 7/19 | 14/51
Other Adverse Events (participants affected / at risk) | 27/28 | 6/6 | 6/6 | 11/11 | 47/48 | 19/19 | 45/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Pooled Placebo 1+2 (N=28) | Part 1: Cohort A: BIIB105 5 mg (N=6) | Part 1: Cohort B: BIIB105 20 mg (N=6) | Part 1: Cohorts C1+C2: BIIB105 60 mg (N=11) | Part 1: Cohorts D1 + D2: BIIB105 120 mg (N=48) | Part 2: BIIB105 60 mg (N=19) | Part 2: BIIB105 120 mg (N=51)
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Pooled Placebo 1+2 (N=28) | Part 1: Cohort A: BIIB105 5 mg (N=6) | Part 1: Cohort B: BIIB105 20 mg (N=6) | Part 1: Cohorts C1+C2: BIIB105 60 mg (N=11) | Part 1: Cohorts D1 + D2: BIIB105 120 mg (N=48) | Part 2: BIIB105 60 mg (N=19) | Part 2: BIIB105 120 mg (N=51)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 7 | 4 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 2 | 3 | 5 | 4 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 4
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 1
Fatigue (General disorders) | 3 | 0 | 0 | 5 | 8 | 3 | 7
Medical device site burn (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 5
Swelling face (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Vaccination site pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 2 | 0 | 0 | 0 | 4 | 4 | 6
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 4
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 3 | 2 | 6
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Stoma site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 3
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 5 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 14 | 1 | 4 | 4 | 18 | 9 | 19
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 2 | 2 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neurological procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 7 | 3 | 1 | 6 | 15 | 7 | 7
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 15 | 5 | 4 | 7 | 25 | 13 | 20
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Shoulder fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 2 | 0 | 3
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 1 | 1 | 3
Stoma site discharge (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Csf protein increased (Investigations) | 0 | 0 | 0 | 0 | 11 | 4 | 7
Csf white blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 6 | 3 | 7
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 4 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 4 | 6 | 3 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3 | 12 | 1 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 1 | 2 | 4 | 3 | 2 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1 | 9 | 3 | 7
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2 | 7 | 2 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 2 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 1 | 0 | 2 | 11 | 4 | 7
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 6 | 0 | 3
Brain fog (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Clonus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cluster headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 2 | 8 | 0 | 5
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 12 | 3 | 4 | 5 | 28 | 5 | 19
Hemihypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Menstrual headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 2 | 0 | 0 | 1 | 2 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleocytosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 6 | 3 | 4
Post-traumatic headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 1
Radicular pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Affect lability (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 3 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 5
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 2 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 3
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Nodular rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 6
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
Study terminated because of sponsor's decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT04494256/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT04494256/SAP_001.pdf